CLINICAL TRIAL: NCT04577612
Title: A Randomized Controlled Test of the Effects of CHI-554 on Fear (F-01)
Brief Title: A Randomized Controlled Test of the Effects of CHI-554 on Fear.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Canopy Growth Corporation (Industry)
Collaborators: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: USA710-4010
Record Dates: First submitted 2020-09-30; First posted 2020-10-08 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Anxiety; Fear; Panic
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Phase 2b, randomized, double-blind, placebo-controlled study
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study. Investigators, study personnel, and participants will be blinded to the group assignment during the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): 150 mg CBD
  Interventions: Drug: CHI-554
- Group 2 (Experimental): 300 mg CBD
  Interventions: Drug: CHI-554
- Group 3 (Experimental): 600 mg CBD
  Interventions: Drug: CHI-554
- Group 4 (Placebo Comparator): Placebo MCT oil
  Interventions: Drug: CHI-554

INTERVENTIONS:
Drug: CHI-554 — hemp-derived CBD in MCT oil

SUMMARY:
This is a randomized, double-blind, placebo-controlled phase 2b clinical trial examining the effects of CHI-554 (CBD) on Fear (F-01)

DETAILED DESCRIPTION:
This study will examine the potential of a novel formulation of hemp-derived CBD (CHI-554) to reduce fear elicited via a safe, well-established, controlled, laboratory-based carbon dioxide (CO2)-enriched air biological challenge that causes abrupt increases in bodily arousal.

ELIGIBILITY:
Inclusion Criteria:

1. Person is between 18 and 55-years-old (inclusive).
2. Person has a BMI between 18 and 35 kg/m2 (inclusive).
3. Person is willing and able to provide informed consent and attend a 3.5-hour, in-person session.
4. Woman of childbearing potential must not be pregnant or currently breastfeeding.
5. If person uses medication, the person has maintained a stable dose and regimen on existing medications for at least 30 days prior to participation in the study and throughout the study.
6. Person agrees to abide by all study restrictions and comply with all study procedures.

Exclusion Criteria:

1. Person has a known history of significant allergic condition, significant hypersensitivity to the IP, or allergic reaction to cannabis, cannabinoid medications, hemp products, or excipients of the IP.
2. Person has been exposed to any investigational drug or device < 30 days prior to screening or plans to take an investigational drug in the near future (within 30 days).
3. Person has used cannabis, synthetic cannabinoid or cannabinoid analogue (e.g., dronabinol, nabilone), synthetic cannabinoid receptor agonist (e.g., spice, K2), or any CBD- or delta-9- tetrahydrocannabinol (THC)-containing product within 30 days of screening or during the study.
4. Person is currently prescribed medications with likely THC- or CBD- interactions (e.g., warfarin, clobazam, valproic acid, phenobarbital, mechanistic target of rapamycin [mTOR] inhibitors, oral tacrolimus, St. John's wort; Epidiolex).
5. Person is currently prescribed and using a medication used in the treatment of anxiety disorders (e.g., selective serotonin uptake inhibitors, venlafaxine, buspirone, benzodiazepines, hydroxyzine, tiagabine, gabapentin, valproate, lamotrigine, topiramate, beta blockers, clonidine, guanfacine, atypical antipsychotics);
6. Person has a positive drug screen for THC, barbiturates, amphetamines, benzodiazepines, and/or opiates at baseline assessment.
7. Person meets diagnostic criteria for a current DSM-5 diagnosis indexed via the MINI.
8. Person meets criteria for a lifetime history of an unexpected or unprovoked panic attack indexed via the MINI.
9. Person endorses current suicidal intent as indexed via the C-SSRS.
10. Person reports a history of being diagnosed with a respiratory or lung disease (including asthma attacks), cardiac or pulmonary disease, epilepsy, narcolepsy, sleep apnea, anemia, or renal disease during a medical history interview.
11. Person has participated in a study that used a CO2-enriched air procedure.
12. Person has received formal training to tolerate elevated levels of CO2 or bodily arousal (such as free diver training or interoceptive exposure-based treatment).
13. Any other clinically significant disease or disorder or abnormal findings during screening or the baseline assessment that, in the opinion of the investigator, may either put the person at risk because of participation in the study, may confound the results of the study, or affect the person's ability to participate in the study.
14. Person has an acute or progressive disease that is likely to interfere with the objectives of the study, or the ability to adhere to protocol requirements.
15. Woman of childbearing potential, unless she has not engaged in vaginal intercourse or she has used effective contraception when doing so (for example, oral contraception, double barrier, intra-uterine device) for at least 30 days prior to the study.
16. Woman of childbearing potential, unless willing to ensure that she or her partner use effective contraception (for example, oral contraception, double barrier, intra-uterine device) during the study and for 30 days thereafter (however, a male condom should not be used in conjunction with a female condom).
17. Man whose partner is of childbearing potential, unless willing to ensure that he or his partner use effective contraception (for example, oral contraception, double barrier, intra-uterine device) during the study and for 30 days thereafter (however, a male condom should not be used in conjunction with a female condom).
18. Person has history of diagnosis related to hepatic function and/or significantly impaired hepatic function (alanine aminotransferase [ALT] >5 ´ upper limit of normal [ULN] or total bilirubin [TBL] >2 ´ ULN) OR the ALT or aspartate aminotransferase (AST) >3 ´ ULN and TBL >2 ´ ULN (or international normalized ratio [INR] >1.5).
19. Person demonstrates behavior indicating unreliability or inability to comply with the requirements of the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Fear ratings | 1 day
  Mean mid-challenge fear ratings measured (via continuous transducer input with a range of 1 to 10, where higher ratings reflect more fear) during seconds 300-330 of the experimental procedure (seconds 150-180 of the biological challenge).

SECONDARY OUTCOMES:
AUC in mean fear ratings | 1 day
  Area under the curve with respect to increase (AUCI) in mean fear ratings (measured via continuous transducer input, with a range of 1 to 10, where higher ratings reflect more fear) sampled at baseline and during 30-second epochs each minute before, during, and after the biological challenge as calculated using the trapezoidal formula.
Self-reported anxiety | 1 day
  Self-reported anxiety (state form of the Spielberger State-Trait Anxiety Inventory (STAI), with a possible range of scores from 20 to80, where higher scores reflect greater anxiety) measured immediately prior to beginning the biological challenge.
AUC in state anxiety ratings | 1 day
  AUC-I in state anxiety ratings (VAS) across the experimental period as calculated using the trapezoidal formula.
Mean intensity using DSQ | 1 day
  mean intensity of physical attack symptoms, cognitive panic attack symptoms, and percentage of participants endorsing a panic attack.

OTHER OUTCOMES:
mean mid-challenge fear ratings | 1 day
  Mean mid-challenge fear ratings (continuous transducer input, with a range of 1 to 10, where higher ratings reflect more fear) during seconds 300-330 of the experimental procedure (seconds 150-180 of the biological challenge) as a function of the interaction between anxiety sensitivity - physical concerns (Physical Concerns sub-scale of the ASI-3) and group (placebo, 150 mg CBD, 300 mg CBD, 600 mg CBD).
mean mid-challenge heart rate | 1 day
  Mean mid-challenge heart rate during seconds 300-330 of the experimental procedure (seconds 150-180 of the biological challenge).
AUC in mean heart rate | 1 day
  AUCI in mean heart rate sampled at baseline and during 30-second epochs each minute before, during, and after the biological challenge as calculated using the trapezoidal formula.
AUC in mean blood oxygen level | 1 day
  AUCI in mean blood oxygen level sampled at baseline and during 30-second epochs each minute before, during, and after the biological challenge as calculated using the trapezoidal formula.

CONTACTS AND LOCATIONS:
Locations (1):
- Ellen W Leen-Feldner, University of Arkansas, Fayetteville, Arkansas, United States